CLINICAL TRIAL: NCT00910039
Title: SUNDANCE Trial: Phase II Trial of Sunitinib as Maintenance Therapy After Stereotactic Radiosurgery in Patients With 1-3 Newly Diagnosed Brain Metastases
Brief Title: Sunitinib Malate After Stereotactic Radiosurgery in Treating Patients With Newly Diagnosed Brain Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1308; P30CA043703 (NIH); CASE1308 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Results first posted 2013-10-01 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Cognitive/Functional Effects; Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: cognitive/functional effects; tumors metastatic to brain; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Sunitinib; Mental Status and Dementia Tests; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib malate (Experimental): Oral sunitinib malate once daily on days 1-28. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Patients undergo neuropsychological battery testing at baseline and periodically during study to assess cognitive function (memory, verbal fluency, visual-motor speed, executive function, and motor dexterity), activities of daily living, and quality of life.
  Interventions: Drug: sunitinib malate; Other: cognitive assessment

INTERVENTIONS:
Drug: sunitinib malate — Treatment will be administered on an outpatient basis. Patients will receive sunitinib 37.5mg once daily in the morning without regard to meals in repeated 6-week cycles comprising daily therapy for 4 weeks followed by a 2-week rest period. Patients who tolerate this dose may increase the dose to 50 mg once daily.
  Other Names: SUNITINIB L-Malate salt; SU010398; PHA-290940AD; Sutent; SUNITINIB
Other: cognitive assessment — The memory test has six alternate forms. The other tests measure motor and information processing speed and are relatively resistant to the effects of practice. The total time for test administration, including the QOL and symptom measures, is 40 minutes.The difference between the pre-treatment baseline and follow-up assessment scores will be determined by the reliable change (RC) index. This index is derived from the standard error of measurement (SEM) for each test in the battery: 1 (deterioration), 2 (no change), or and 3 (improved).
  Other Names: Cognitive Function Tests:; Memory Hopkins Verbal Learning Test; Verbal fluency Controlled Oral Word Association; Visual-motor speed Trail Making Test Part A; Executive Function Trail Making Test Part B; Motor dexterity Grooved Pegboard 3; Function Test:; Quality of life (QOL) was evaluated with a self-report measure (FACT-BRREF).

SUMMARY:
RATIONALE: Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sunitinib malate works after stereotactic radiosurgery in treating patients with newly diagnosed brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the CNS progression-free survival rate in patients with 1-3 newly diagnosed brain metastases treated with sunitinib malate after stereotactic radiosurgery (SRS).

Secondary

* Determine the rate of local (site of SRS treatment) failure at 12 months in these patients.
* Determine the median time to CNS disease progression in these patients.
* Determine the overall survival of these patients.
* Determine the time to progression of systemic disease in these patients.
* Evaluate the safety of sunitinib malate when administered after SRS in these patients.
* Assess the neurocognitive effects of SRS followed by sunitinib malate in these patients.

OUTLINE: Patients receive oral sunitinib malate once daily on days 1-28. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.

Patients undergo neuropsychological battery testing at baseline and periodically during study to assess cognitive function (memory, verbal fluency, visual-motor speed, executive function, and motor dexterity), activities of daily living, and quality of life.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed carcinoma
* Has 1-3 newly diagnosed brain metastases amenable to stereotactic radiosurgery
* Patients may enroll up to 1 month after the completion of stereotactic radiosurgery provided they can undergo the required neuropsychiatric battery before beginning treatment.
* Patients must begin treatment within 1 month of stereotactic radiosurgery.
* No CNS metastases from lymphoma or small cell lung cancer
* No leptomeningeal metastases
* No CNS complications requiring urgent neurosurgical intervention (e.g., resection or shunt placement)

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100% (RTOG RPA class I or II)
* Life expectancy > 6 weeks
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL (transfusion allowed)
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Total serum bilirubin ≤ 1.5 times ULN
* Serum calcium ≤ 12.0 mg/dL
* Serum creatinine ≤ 2.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing and able to comply with schedule visits, treatment plans, laboratory tests, and other study procedures
* No medical problem (unrelated to the malignancy) that would pose an undue risk or that would limit full compliance with the study
* No unresolved bowel obstruction
* No uncontrolled infectious process
* No evidence of bleeding diathesis or coagulopathy

  * Hematuria from a primary renal tumor is allowed provided all other eligibility criteria are met
* No hypertension that cannot be controlled by medications to a blood pressure of < 160/90 mm Hg
* None of the following within the past 6 months:

  * Myocardial infarction
  * Severe/unstable angina
  * Severe peripheral vascular disease (claudication) or procedure on peripheral vasculature
  * Coronary/peripheral artery bypass graft
  * NYHA class II-IV congestive heart failure
  * Cerebrovascular accident or transient ischemic attack
  * Clinically significant bleeding
  * Deep venous thrombosis or pulmonary embolism
* No other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or that may interfere with the interpretation of study results and, in the judgement of the investigator, would make the patient inappropriate for entry into this study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior sunitinib malate
* No prior cranial external beam radiotherapy
* No concurrent coumadin or other agents containing warfarin, except for low-dose coumadin (≤ 1 mg) administered prophylactically for maintenance of in-dwelling lines or ports
* No concurrent hepatic enzyme-inducing anticonvulsants
* No concurrent participation in another clinical trial
* No other concurrent investigational agents
* Concurrent steroids allowed provided dose is stable for ≥ 1 week
* Concurrent systemic therapy for management of stable systemic disease allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-04; Primary Completion 2012-01 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M. Peereboom, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Henry Ford Health System, Detroit, Michigan
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fourteen patients were entered onto this trial between 8/2009 and 6/2011 from Cleveland Clinic and Henry Ford Health System.
Groups:
- Sunitinib Malate: Oral sunitinib malate (37.5mg) once daily on days 1-28. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Patients undergo neuropsychological battery testing at baseline and periodically during study to assess cognitive function (memory, verbal fluency, visual-motor speed, executive function, and motor dexterity), activities of daily living, and quality of life.
Period: Overall Study
Arm/Group | Sunitinib Malate
Started | 14
Completed | 13
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Sunitinib Malate: Oral sunitinib malate (37.5mg)once daily on days 1-28. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Patients undergo neuropsychological battery testing at baseline and periodically during study to assess cognitive function (memory, verbal fluency, visual-motor speed, executive function, and motor dexterity), activities of daily living, and quality of life.
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 59 [46 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Central Nervous System (CNS) Progression-free Survival Rate
Description: The number of subjects surviving at least six months from SRS without progressive disease anywhere in the brain (local or regional failure), assessed by the McDonald's standard criteria.Progressive neurologic abnormalities not explained by causes unrelated to tumor progression (e.g. anticonvulsant or corticosteroid toxicity, electrolyte abnormalities, hyperglycemia, etc.) or a greater than 25% increase in the size of the tumor by MRI/CT scan.
Time Frame: 6 months after stereotactic radiosurgery (SRS)
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 14
participants | 7 [37 to 63]

2. Secondary Outcome: Central Nervous System (CNS) Progression-free Survival Rate
Description: The number of subjects surviving at least 12 months from SRS without progressive disease anywhere in the brain (local or regional failure), assessed by the McDonald's standard criteria. Progressive neurologic abnormalities not explained by causes unrelated to tumor progression (e.g. anticonvulsant or corticosteroid toxicity, electrolyte abnormalities, hyperglycemia, etc.) or a greater than 25% increase in the size of the tumor by MRI/CT scan.
Time Frame: 12 months after stereotactic radiosurgery (SRS)
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 14
participants | 6

3. Secondary Outcome: Median Time to CNS Disease Progression
Description: Time to disease progression will be recorded from the first day of protocol therapy until the criteria for disease progression are met, patient death from any cause or removal of the patient from study for any reason, whichever comes first.
Time Frame: up to12 months from SRS
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 14
months | 6.6 [1.5 to 19]

4. Secondary Outcome: Overall Survival
Description: The number of subjects surviving at least 12 months from stereotactic radiosurgery.
Time Frame: 12 months from SRS
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 14
participants | 7

5. Secondary Outcome: Time to Progression
Description: Time to progression (all sites of disease) - interval between stereotactic radiosurgery and the earliest date of progression (systemic or CNS) or death due to any cause.
Time Frame: at 3 yrs from SRS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 14
months | 4.8 [1.5 to 18.8]

6. Secondary Outcome: Rate of Local Failure at 12 Months
Description: Rate of local vs regional failure -rates of progression at site of stereotactic radiosurgery (local failure)vs progression anywhere else in CNS (regional failure).
Time Frame: 12 months
Population: Due to the small number of patients accrued there was not enough data for analysis of this outcome.
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 0

7. Secondary Outcome: Neurocognitive Effects
Description: The number of patients that had statistically significant change (p's > 0.05) in their neurocognitive assessment (improvement or decline) from baseline. Neurocognitive function was assessed in several domains, including memory, verbal fluency, visual-motor speed, executive function and motor dexterity.The difference between the pre-treatment baseline and follow-up assessment scores were determined by the reliable change (RC) index. RC Index: 1=deterioration, 2=no change, 3=improved
Time Frame: at 2 months after treatment
Population: Due to the small number of patients accrued there was not enough data for analysis of this outcome.
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 0

8. Secondary Outcome: Safety and Tolerability
Description: Number of patients that experienced treatment-related G 3-4 adverse events.
Time Frame: 3 years from study start
Measure: Number; unit: participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 14
participants | 9

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from on study date to off study for a period of about 2.5 years.
Arm/Group | Sunitinib Malate
Serious Adverse Events (participants affected / at risk) | 7/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib Malate (N=14)
Lymphopenia (Blood and lymphatic system disorders) | 2
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1
Cardiac troponin T (cTnT) (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Hemorrhage, CNS (Nervous system disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 1
Aphasia (Nervous system disorders) | 1
Pain - Head/headache (Nervous system disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib Malate (N=14)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 3
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 5
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3
Platelets (Blood and lymphatic system disorders) | 7
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 2
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 1
INR (International Normalized Ratio of prothrombin time) (Investigations) | 1
Lightheadedness (Nervous system disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 14
Insomnia (Psychiatric disorders) | 2
Rigors/chills (General disorders) | 1
Weight gain (Investigations) | 1
Weight loss (Investigations) | 1
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1
Icteric Skin (Jaundice) (Skin and subcutaneous tissue disorders) | 2
Dermatology/Skin - Other (NOS) (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 6
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 10
Heartburn/dyspepsia (Gastrointestinal disorders) | 3
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 6
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 6
Hemorrhage, pulmonary/upper respiratory - Lung (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1
Sub-conjunctival hemorrhage (Eye disorders) | 1
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - External ear (otitis externa) (Ear and labyrinth disorders) | 1
Edema: limb (General disorders) | 4
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 5
Albumin, serum-low (hypoalbuminemia) (Investigations) | 1
Calcium, serum-high (hypercalcemia) (Investigations) | 2
Creatinine (Investigations) | 4
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1
Proteinuria (Metabolism and nutrition disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 1
Confusion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Mood alteration - Agitation (Nervous system disorders) | 2
Mood alteration - Anxiety (Nervous system disorders) | 2
Mood alteration - Depression (Nervous system disorders) | 2
Neurology - Other (Right-sided Facial Drooping) (Nervous system disorders) | 1
Neurology - Other (Shaking, right leg and arm) (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 1
Speech impairment (Slurred Speech) (Nervous system disorders) | 1
Syncope (fainting) (Nervous system disorders) | 1
Eye twitching (Nervous system disorders) | 1
Vision-blurred vision (Eye disorders) | 1
Watery eye (epiphora, tearing) (Eye disorders) | 1
Pain - Abdominal cramps (Gastrointestinal disorders) | 2
Pain - Back (Musculoskeletal and connective tissue disorders) | 2
Pain - Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 1
Pain - External ear (Musculoskeletal and connective tissue disorders) | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 2
Pain - Head/headache (Nervous system disorders) | 5
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1
Pain - Jaw (Musculoskeletal and connective tissue disorders) | 1
Pain - Other (left groin pain) (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1
Obstruction, GU - Ureter (Renal and urinary disorders) | 1
Obstruction, GU - Urethra (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes